CLINICAL TRIAL: NCT01744327
Title: An Exploratory Study Investigating TL1A Expression in Psoriatic Skin and Serum and Monocytes Capacity to Produce TL1A
Brief Title: TL1A Expression in Psoriatic Skin
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: AbbVie (Industry); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Bo Bang, MD, Ph.D, Chief Physician, Associate Professor, Bispebjerg Hospital
Other Study IDs: 331536
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Plaque type psoriasis: Patients with plaque type psoriasis

SUMMARY:
TL1A is a newly discovered signal molecule that may be crucially involved in the maintenance of chronic inflammatory disorders. TL1A has also been demonstrated in psoriatic skin but the importance of TL1A in psoriasis is still unknown. Understanding inflammatory signal molecules in psoriasis is important because the development of new drugs directed against relevant signal molecules (e.g. TNF-α and IL12/23) has proved to be a very efficacious treatment principle. However, despite the dramatic progress in therapeutic options during the last decade, there is still a fraction of patients that are insufficiently treated with the currently available therapies. TL1A has been claimed to be the next important target for development of biologics in the field of chronic inflammation.

DETAILED DESCRIPTION:
Psoriasis is a common autoimmune disease; affecting approximately 2 % of the western population. Among these 15% are estimated to have severe disease that requires systemic therapy with e.g. methotrexate, cyclosporine or acitretin that are all drugs associated with high frequencies of side-effects. In contrast to this the recent development of the biologic drugs has provided very efficacious and in general well-tolerated new therapeutics. But even with these newer drugs treatment-failures exist and for this group new treatments are needed TNF-like ligand 1A (TL1A) is a novel member of the TNF family of cytokines. Increasing evidence suggests that in addition to TNF-alfa and IFN-gamma psoriasis is also an IL-23 and IL-17 dependent disease so TH1 and TH17 T cells are suggested to be important in driving the disease. Therefore TL1A, which through binding to DR3 influences TH1 and TH17 T cell differentiation, could be an important cytokine in the early inflammatory process in psoriasis. Recently expression of TL1A in psoriatic skin lesions has been demonstrated but the importance of this remains to be investigated.

TL1A exists in both a membrane bound- and a soluble form and is secreted from antigen presenting cells (APCs) such as monocytes, dendritic cells and macrophages in response to stimulation with immune complexes, bacteria or cytokines (TNF-alfa and IL-1beta). Membrane bound TL1A has also been described in T cells. Recently, a new isoform of soluble TL1A (TL1A(V84-L251)) was discovered with functional differences to TL1A(L72-L251. It's unknown whether this isoform is present in psoriatic skin.

Research on TL1A has focused on autoimmune diseases where immune complexes are formed, e.g. rheumatoid arthritis. However, studies have suggested that early pathogenesis in psoriasis could dependent on formation of large complexes between bacterial DNA and the anti-microbial peptide LL-37 which induce cytokine secretion from APC. Cytokines that could lead to TL1A excretion. Whether TL1A can be secreted in this way is unknown.

ELIGIBILITY:
Inclusion Criteria:

* Plaque type psoriasis
* at least 6 month history of psoriasis

Exclusion Criteria:

* systemic anti-psoriatic medication
* topical anti-psoriatic medication (wash-out period 2 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Plaque type psoriasis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Expression of TL1A in psoriatic skin | 3 months
  Staining intensity of TL1A by IHC in involved psoriatic skin compared to uninvolved and skin from normal controls

CONTACTS AND LOCATIONS:
Locations (1):
- Department of dermatology D40 , Bispebjerg Hospital, Copenhagen, Denmark